CLINICAL TRIAL: NCT02703649
Title: Administration of Single High Dose Letrozole for Ovulation Induction - A Randomized Controlled Trial
Brief Title: Administration of Single High Dose Letrozole for Ovulation Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Siba0101
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Anovulation
Keywords: Aromatase inhibitor; induction of ovulation
MeSH Terms: conditions — Anovulation | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single dose (Experimental): Single 20 mg dose of Letrozole on day 3 of the menstrual cycle.
  Interventions: Drug: Letrozole
- Daily dose (Active Comparator): Daily dose of Letrozole 2.5 mg starting day 3 for 5 days.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — After the decision to use Letrozole for induction of ovulation, we will obtain informed consent and randomize the patents into 2 groups Single 20 mg dose of Letrozole on day 3 of the cycle Daily dose of Letrozole 2.5 mg starting day 3 for 5 days.
  Other Names: Femara

SUMMARY:
Letrozole is considered an established treatment for ovulation induction.The most common protocol is daily dose of 2.5-7.5 mg starting day 3-5 of the cycle for 5 days.Another described protocol is single high dose 20mg Letrozole given on day 3 of the cycle.

Our aim is to compare the single high dose Letrozole protocol to daily low dose protocol.

DETAILED DESCRIPTION:
Pre-study screening will be conducted before the enrolment in the study, routine fertility assessment: Physical history including fertility and fertility treatment history. Laboratory tests-cycle day 3 hormonal profile (Estradiol, Luteinizing hormone, Follicular stimulating hormone, progesterone), cycle day 3 antral follicular count.

Pregnancy will be excluded by Human chorionic gonadotropin test at day 3 of the cycle, before starting the fertility treatment.

Polycystic syndrome (PCOS) patients will be defined according to Rotterdam criteria 2003.

A prospective randomized clinical trial. PCOS patients who require induction of ovulation will prospectively randomized into two groups:

1. Single 20 mg dose of Letrozole on day 3 of the menstrual cycle. Monitoring for response will include the usual measurements of serum Estradiol (E2), Follicle stimulating hormone (FSH), Luteinizing Hormone (LH), Progesterone (P) and transvaginal ultrasound for follicular count and endometrial thickness measurement. First monitoring will be on day 7 of the cycle and the rest of the monitoring will be determined according to response.
2. Daily dose of Letrozole 2.5 mg starting day 3 for 5 days. Monitoring for response will include serum Estradiol (E2), Follicule stimulating hormone (FSH), Luteinizing Hormone (LH ), Progesterone (P) and transvaginal ultrasound for follicular count and endometrial thickness measurement. First day of monitoring will be on day 7 and the rest of monitoring will be determined according to response.

Statistical Analysis

* Primary Endpoint Analysis: Sample Size Selection In order to prove non-inferiority with significance level (alpha) 5% and power of 90%, standard deviation of outcome 1, and noninferiority limit 1; the sample size needed is 36 patients in both groups. Calculation based on Jolious SA formula.(7)
* Planned Analysis

Primary Outcome Analysis:

Comparison of the number of follicle >15 mm at day of ovulation

Secondary Outcome Analysis:

Pregnancy rate Comparison between the two groups Estradiol levels at day of ovulation triggering Ovarian hyperstimulation syndrome Clinical pregnancy rate

Statistical analysis :

The various outcome measures will be expressed as numbers and rates. The Student t test, χ2 test and analysis of variance will be used where appropriate to analyze the various data among the study groups. P value less than .05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (PCOS) patients
* BMI (body mass index) of 18-35.
* Proved one patent fallopian tube at least

Exclusion Criteria:

* Women with low ovarian response (According to Bologna criteria )
* Blocked fallopian tubes
* Pregnancy
* Presence of any clinically significant health problem such that treatment with letrozole or pregnancy would not be in the subject's best interest.
* Co-administration of other anti-estrogens
* Hypersensitivity to Letrozole .

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03; Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
number of follicles >15 mm at day of ovulation | First day of monitoring will be on day 7 and the rest of monitoring will be appointed according to response up to 1month

SECONDARY OUTCOMES:
Pregnancy rate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Casper, MD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, University of Toronto, Toronto, Ontario
  - TRIO Fertility, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franik S, Le QK, Kremer JA, Kiesel L, Farquhar C. Aromatase inhibitors (letrozole) for ovulation induction in infertile women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2022 Sep 27;9(9):CD010287. doi: 10.1002/14651858.CD010287.pub4. PMID 36165742